CLINICAL TRIAL: NCT04799964
Title: Efficacy and Safety of the Flow Diverter (Tonbridge) for Endovascular Treatment of Intracranial Aneurysms: a Prospective, Multi-center, Randomized, Open, Positive-controlled, Non-inferiority Trial
Brief Title: Efficacy and Safety of the Flow Diverter (Tonbridge) for Endovascular Treatment of Intracranial Aneurysms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ton-Bridge Medical Tech. Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZHTQ2020001
Record Dates: First submitted 2021-02-20; First posted 2021-03-16 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Flow Diverter (Tonbridge) (Experimental): Treatment with Flow Diverter (Tonbridge)
  Interventions: Device: Flow Diverter (Tonbridge)
- Tubridge (MicroPort) (Active Comparator): Treatment with Tubridge (MicroPort)
  Interventions: Device: Tubridge (MicroPort)

INTERVENTIONS:
Device: Flow Diverter (Tonbridge) — The device is a self-expanding vascular stent system, which consists of a stent and a delivery system. The stent is made of platinum core nickel-titanium alloy material. The delivery system is composed of a delivery guide wire and an introducer sheath. The stent and the delivery guide wire are pre-installed in the introducer sheath.
  Arms: Flow Diverter (Tonbridge)
Device: Tubridge (MicroPort) — Tubridge consists of a stent system and a microcatheter system. The stent system consists of a stent and a conveyor, the stent is self-expanding as well.
  Arms: Tubridge (MicroPort)

SUMMARY:
The purpose of this study is to assess the efficacy and safety of the Flow Diverter (Tonbridge) for endovascular treatment of intracranial aneurysms.

DETAILED DESCRIPTION:
This is a prospective, multi-center, randomized, open, positive-controlled, non-inferiority trial. This clinical trial is conducted at more than 5 centers in China. Eligible patients are randomized into experimental group using Flow Diverter (Tonbridge) or control group using Tubridge (MicroPort) in a 1:1 ratio. The primary objective of this study is to verify the complete occlusion rate of aneurysms at 12 months of Flow Diverter (Tonbridge) is non-inferior to Tubridge, for treatment of intracranial aneurysms, and evaluate the effectiveness and safety of the Flow Diverter (Tonbridge).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years, any gender;
* Unruptured intracranial aneurysms locate in the internal carotid artery (ICA) or vertebral artery (VA) with a neck ≥ 4 mm and a maximal diameter ≥ 10 mm, which diagnosed by DSA;
* The target aneurysm with a parent vessel diameter of 2.0-6.5 mm;
* Subject or guardian is able to understand the purpose of study, shows sufficient compliance with the study protocol and provides a signed informed consent form.

Exclusion Criteria:

* Diagnosed as multiple aneurysms which cannot be covered by a single stent or with cerebrovascular malformations;
* Subarachnoid hemorrhage of the target aneurysm within 30 days pre-procedure;
* Modified Rankin Scale (mRS) score > 2 in pre-procedure;
* Platelet (PLT) < 60×10^9/L or known platelet dysfunction or International Normalized Ratio (INR) > 1.5;
* Heart, lung, liver and renal failure or other severe diseases (such as brain tumor, systemic infection, disseminated intravascular coagulation, myocardial infarction within 12 months before enrollment, history of severe psychosis);
* The lesion which is not appropriate for flow diverter delivery and deployment judged by investigators (severe stenosis of parent artery, severe tortuosity of parent artery, stent failing to reach the lesion, etc.);
* Major surgery within 30 days before enrollment, or intending to receive surgery within 180 days after enrollment;
* Allergic history of anesthetics and contrast agents, or contraindication for dual antiplatelet or/and anticoagulant therapy;
* Allergic History of metals such as nickel-titanium alloy;
* Life expectancy < 12 months;
* Pregnant or breastfeeding women;
* Subject has participated in other drug or medical device clinical trials within 1 month before signing informed consent;
* Other conditions judged by the investigators as unsuitable for enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Complete occlusion rate of aneurysms at 12 months | 360±45 days post-procedure
  Complete occlusion is defined as no contrast agent in the aneurysm (Raymond-Roy class I) which is diagnosed by cerebrovascular DSA at 12 months post-procedure.

SECONDARY OUTCOMES:
Immediate procedural success rate | intra-procedure
  Intraoperative cerebrovascular DSA is performed to determine whether the investigational device positions exactly and covers the aneurysm neck effectively.
Complete occlusion rate of aneurysms at 6 months | 180±30 days post-procedure
  Complete occlusion is defined as no contrast agent in the aneurysm (Raymond-Roy class I) which is diagnosed by MRA/CTA at 6 months post-procedure.
Subtotal occlusion rate | 360±45 days post-procedure
  Subtotal occlusion is defined as contrast agents in the aneurysm sac less than 10% which is diagnosed by DSA at 12 months post-procedure.
Incidence of technical complications | intra-procedure
  Technical complications include but not limited to: stent incomplete opening, stent migration, stent herniation into the aneurysm sac, in-stent thrombosis, operation injury, etc.
Incidence of stroke | within 360±45 days
  Stroke includes hemorrhagic stroke and symptomatic ischemic stroke.
Incidence of parent artery stenosis ( > 50%) in target area at 360 days and incidence of parent artery occlusion in target area at 360 days | 360±45 days post-procedure
  Parent artery stenosis in target area is defined as stenosis degree > 50%. Using postoperative cerebrovascular DSA at 360 days is performed to determine.
Incidence of adverse events and incidence of serious adverse events | within 360±45 days
  "Incidence of adverse events" is the proportion of subjects with adverse events using the investigational device or the comparator;
  "Incidence of serious adverse events" is the proportion of subjects with serious adverse events using the investigational device or the comparator.
Mortality rate | within 360±45 days
  Deaths due to any cause are calculated.
Operation satisfaction rate | intra-procedure
  The 5-point Likert scale is used to evaluate the operation satisfaction from three aspects: push performance, retracting performance and release performance. "Operation satisfaction rate" is defined as the proportion of investigational devices or comparators with Likert score ≥ 12 points.
Incidence of device deficiency | within 360±45 days
  Device deficiency is the unreasonable risk that may endanger human health and life safety in the normal use of medical devices during clinical trials, such as labeling errors, quality problems, malfunctions, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Liu, Principal Investigator — Changhai Hospital
Locations (13):
- China (13):
  - The First Affiliated Hospital of USTC, Hefei, Anhui
  - Nanfang Hospital Southern Medical University, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Nanyang Central Hospital, Nanyang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Yichang Central People's Hospital, Yichang, Hubei
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Hospital, Hangzhou, Zhejiang
  - Changhai Hospital of Shanghai, Shanghai
  - Huashan Hospital Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No